CLINICAL TRIAL: NCT04041791
Title: Supportive Care and Antibiotics for Severe Pneumonia Among Hospitalized Children (SEARCH): A Pragmatic Randomised Controlled Trial
Brief Title: A Study to Compare Different Antibiotics and Different Modes of Fluid Treatment for Children With Severe Pneumonia
Acronym: SEARCH
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: University of Nairobi (Other); London School of Hygiene and Tropical Medicine (Other); National Institute for Health Research, United Kingdom (Other Government); Department for International Development, United Kingdom (Other Government); Medical Research Council (Other Government); Wellcome Trust (Other); Kenya Ministry of Health (Other Government)
Responsible Party: Principal Investigator, Ambrose Agweyu, Principal Investigator, University of Oxford
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: KEMRI/CGMR-C/141/3772
Record Dates: First submitted 2019-07-29; First posted 2019-08-01 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Pneumonia
Keywords: severe pneumonia; supportive care; antibiotics; World Health Organisation; intravenous fluids; nutrition; children
MeSH Terms: conditions — Pneumonia | interventions — Penicillin G; Gentamicins; Ceftriaxone; Amoxicillin-Potassium Clavulanate Combination; Ringer's Lactate; Glucose; Saline Solution; Ampicillin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Benzyl penicillin/ampicillin + gentamicin & IV fluids (Active Comparator): Participants are assigned to receive benzyl penicillin at 50,000 IU/kg every 6 hours or ampicillin 50mg/kg every 8 hours plus gentamicin 7.5 mg/kg once daily given intravenously (IV) or via intramuscular (IM) injection for a minimum of 48 hours and for up to 7 days.
  Maintenance fluids will be given as a continuous infusion for at least 24 hours.
  Interventions: Drug: Benzyl penicillin; Drug: Gentamicin Sulfate; Other: Intravenous fluid; Drug: Ampicillin
- Ceftriaxone and IV fluids (Experimental): Participants are assigned to receive ceftriaxone at 50 mg/kg every 12 hours given IV or IM for a minimum of 48 hours and for up to 7 days.
  Intravenous fluids will be given as a continuous infusion for at least 24 hours.
  Interventions: Drug: Ceftriaxone; Other: Intravenous fluid
- Amoxicillin-clavulanate and IV fluids (Experimental): Participants are assigned to receive amoxicillin clavulanic acid at 30 mg/kg every 8 hours given IV or IM for a minimum of 48 hours and for up to 7 days.
  Intravenous fluids will be given as a continuous infusion for at least 24 hours.
  Interventions: Drug: Amoxicillin Clavulanate; Other: Intravenous fluid
- Benzyl penicillin/ampicillin + gentamicin & NG feeds (Experimental): Participants are assigned to receive Benzyl penicillin at 50,000 IU/kg every 6 hours or ampicillin 50mg/kg every 8 hours plus gentamicin 7.5 mg/kg once daily given intravenously (IV) or via intramuscular (IM) injection for a minimum of 48 hours and for up to 7 days.
  Nasogastric feeds will be given 3 hourly for at least 24 hours.
  Interventions: Drug: Benzyl penicillin; Drug: Gentamicin Sulfate; Other: Nasogastric feeds; Drug: Ampicillin
- Ceftriaxone and NG feeds (Experimental): Participants are assigned to receive ceftriaxone at 50 mg/kg every 12 hours given IV or IM for up to 7 days.
  Nasogastric feeds will be given 3 hourly for at least 24 hours.
  Interventions: Drug: Ceftriaxone; Other: Nasogastric feeds
- Amoxicillin-clavulanic acid and NG feeds (Experimental): Participants are assigned to receive amoxicillin clavulanic acid at 30 mg/kg every 8 hours given IV or IM for up to 7 days.
  Nasogastric feeds will be given 3 hourly for at least 24 hours.
  Interventions: Drug: Amoxicillin Clavulanate; Other: Nasogastric feeds

INTERVENTIONS:
Drug: Benzyl penicillin — Benzyl penicillin is a penicillin antibiotic.
  Other Names: Medipen; Cristapen
  Arms: Benzyl penicillin/ampicillin + gentamicin & IV fluids; Benzyl penicillin/ampicillin + gentamicin & NG feeds
Drug: Gentamicin Sulfate — Gentamicin is an aminoglycoside antibiotic.
  Other Names: Gentamicin; Gentamed
  Arms: Benzyl penicillin/ampicillin + gentamicin & IV fluids; Benzyl penicillin/ampicillin + gentamicin & NG feeds
Drug: Ceftriaxone — Ceftriaxone is a third generation cephalosporin antibiotic active against a wide range of gram negative and positive bacteria.
  Other Names: Desefin
  Arms: Ceftriaxone and IV fluids; Ceftriaxone and NG feeds
Drug: Amoxicillin Clavulanate — Amoxicillin Clavulanate is a combination of amoxicillin, a β-lactam antibiotic, and potassium clavulanate, a β-lactamase inhibitor.
  Other Names: Amoxicillin-clavulanic acid; Amoxi-clav; Amoklavin; Co-amoxiclav
  Arms: Amoxicillin-clavulanate and IV fluids; Amoxicillin-clavulanic acid and NG feeds
Other: Intravenous fluid — Maintenance fluids administered for at least 24 hours.
  Other Names: Hartmann's Solution with 5% dextrose; Ringer's Lactate with 5% dextrose; Normal Saline with 5% dextrose
  Arms: Amoxicillin-clavulanate and IV fluids; Benzyl penicillin/ampicillin + gentamicin & IV fluids; Ceftriaxone and IV fluids
Other: Nasogastric feeds — Feeds given via nasogastric tube. Feeds may include cow's milk, breast milk, porridge, formula among others.
  Arms: Amoxicillin-clavulanic acid and NG feeds; Benzyl penicillin/ampicillin + gentamicin & NG feeds; Ceftriaxone and NG feeds
Drug: Ampicillin — Ampicillin is a penicillin-type antibiotic.
  Arms: Benzyl penicillin/ampicillin + gentamicin & IV fluids; Benzyl penicillin/ampicillin + gentamicin & NG feeds

SUMMARY:
Pneumonia is one of the top causes of death in children aged below 5. More than 10% of children with severe pneumonia die. We are not sure that the currently recommended antibiotics used in children with pneumonia are the most effective. No studies have been carried out to find out whether children with pneumonia should be given intravenous (IV) fluids or nasogastric (NG) feeds.

The SEARCH trial aims to find out which antibiotics and modes of feeding are the most effective in treating children with severe pneumonia and therefore helping reduce mortality.

DETAILED DESCRIPTION:
Pneumonia is one of the leading causes of death among young children with more than 10% of children aged under-five with severe pneumonia dying. The World Health Organisation (WHO) guidelines recommend the use of benzyl penicillin plus gentamicin as the standard of care of treatment for severe pneumonia. However, there have been increasing concerns about the effectiveness of the current recommendations.

Some authorities advise against the use of enteral nutrition in severely ill patients due to concerns of compromised respiratory status and risk of aspiration with nasogastric feeding. Evidence to support these concerns is lacking.

This trial aims to find out which antibiotics are the most effective in the treatment of children with severe pneumonia by comparing the current standard of care (benzyl penicillin or ampicillin plus gentamicin) to injectable ceftriaxone and injectable amoxicillin-clavulanic acid. The study will also determine whether providing feeds through a nasogastric tube is superior to intravenous fluid therapy in children with severe pneumonia.

The SEARCH trial will be a multi-site pragmatic randomised controlled trial that will assess the efficacy of both interventions in children admitted with severe pneumonia in a 3x2 factorial design. The sites will be in East Africa.

Data from the trial will be used to inform policy and contribute to guidelines and improve clinical practice in settings where the burden of pneumonia is highest.

ELIGIBILITY:
Inclusion Criteria:

* Age 2 to 59 months.
* History of cough or difficulty breathing and signs of severe pneumonia based on WHO 2013 criteria
* Admitted to any one of the study hospitals.
* Informed consent provided by the parents/guardian.

Exclusion Criteria:

* Children presenting in cardiorespiratory arrest requiring emergency basic life support (bag-valve-mask ventilation and/or chest compressions).
* Children for whom concurrent condition precludes the use of the first-line antibiotics for severe pneumonia such as readmission or meningitis
* Known allergy or contraindication to penicillin, gentamicin, ceftriaxone or amoxicillin-clavulanic acid.
* Referral from another inpatient facility following treatment with injectable antibiotics for more than 24 hours or because the first-line regimen is considered to have failed
* Previously enrolled in the study.
* For supportive care intervention (Intravenous fluids versus nasogastric feeds): children with absent gag reflex.
* For supportive care intervention (Intravenous fluids versus nasogastric feeds): children unable to maintain oxygen saturations greater 90% on pulse oximetry while receiving supplemental oxygen.
* For supportive care intervention (Intravenous fluids versus nasogastric feeds): children with severe acute malnutrition
* For supportive care intervention (Intravenous fluids versus nasogastric feeds): shock or severe dehydration
* For supportive care intervention (Intravenous fluids versus nasogastric feeds): Child able to feed
* For supportive care intervention (Intravenous fluids versus nasogastric feeds): Vomiting everything

Ages: 2 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 4392 (Actual)
Dates: Start 2019-08-19 (Actual); Primary Completion 2024-04-05 (Actual); Study Completion 2024-04-05 (Actual)

PRIMARY OUTCOMES:
Mortality | Up to Day 5
  Mortality of participants receiving any of the injectable antibiotic treatments who die within the first five days of admission measured from source documents, medical records, verbal autopsy or death certificates.

SECONDARY OUTCOMES:
Number of serious adverse events | Up to Day 30
  Serious adverse events that my be likely or definitely related to any of the interventions given to the participants. Serious adverse events include death, a life threatening event, persistent or significant disability or incapacity, hospitalisation or prolonged hospitalisation.
Length of hospitalisation | Through duration of hospitalisation, an average of 5 days
  Total days a participant is admitted or receives inpatient care measured in days using hospital records at the start and end of each admission.
Duration taken to tolerate full fluids by mouth | An average of 3 days
  Number of days it takes for participants to fully tolerate fluids orally.
Mortality 30 days after enrollment | Day 30 post enrollment
  Number of participants who die within 30 days of enrollment into the study measured using source documents, medical records, verbal autopsy or death certificates.

CONTACTS AND LOCATIONS:
Overall Officials: Ambrose Agweyu, PhD, Principal Investigator — KEMRI-Wellcome Trust Research Programme, University of Oxford
Locations (1):
- Machakos Level 5 Hospital, Machakos, Kenya

IPD SHARING:
Plan to Share IPD: No
Data requests will be considered by applying to the Data Governance Committee at the Kenya Medical Research Institute (KEMRI) Centre for Geographic Medicine Research-Kilifi, Kenya who will manage the process and ensure that appropriate ethical approval is in place and consent has been obtained for dissemination and use outside of the scope of the trial.